CLINICAL TRIAL: NCT04581642
Title: Nociception-Level (NOL) for the Assessment of Pain in Patient Unable to Self-Report: An Exploratory, Prospective, Unblinded, Single-center Study- The MoNOLog Study
Brief Title: Nociception-Level (NOL) for the Assessment of Pain in Patient Unable to Self-Report
Acronym: MoNOLog
Status: Completed | Type: Observational
Sponsor: Medasense Biometrics Ltd (Other)
Responsible Party: Sponsor
Other Study IDs: CLI-01-1-09
Record Dates: First submitted 2020-10-03; First posted 2020-10-09 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Pain; Opioid Use; Dementia; Unconscious; Ventilator Lung
MeSH Terms: conditions — Pain; Dementia; Unconsciousness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: PMD200 — The NOL technology is comprised of a console and designated finger probe with 4 sensors. The Sensors are Photoplethysmography (PPG) Galvanic Skin Response (GSR), Accelerometer (ACC) and Thermistor (TMP)

SUMMARY:
In this study we aimed to investigate the performance and effectiveness of NOL and/or NOLedge as a tool for pain assessment in geriatric and critical ill non communicating patients.

Our hypothesis was that NOL and the NOLedge may have good correlation with the health-care professional assessment PAINAD, BPS values, even with the use of the drugs affecting autonomic nervous system.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, Age > 18 years old.
* Spontaneously breathing or mechanically ventilated
* Any patient who is unable to express his/her own level of personal pain by using visual scales according to the hospital standard
* Written informed consent provided by the participant (if they have capacity) or guardian (if they do not have capacity) or a written proxy informed consent from a legally authorized representative empowered to make health-related decisions for the potential study participant.

Exclusion Criteria:

* A patient whose staff or research team believes that his or her participation in the research will cause suffering to the patient.
* Unstable condition preventing planned routine procedures of care, and conditions precluding the use of PMD-200: absence of sinus cardiac rhythm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a clinical syndrome due to disease of a progressive nature, which leads to disturbances in multiple higher cortical functions, including memory, thinking, orientation, comprehension, calculation, learning capacity, language and judgment;
  1. Older adults with advanced dementia;
  2. Critically ill/unconscious patients;
  3. Patients at the end of life stage.
  4. Ventilated patients.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Efficacy outcome | 5 months
  To identify what information is currently elicited and used by clinicians when detecting and managing pain.
Efficacy outcome | 5 months
  To assess the feasibility of the current NOL algorithm (PMD200 vs. NOLedge) for pain management in the study population.
Efficacy outcome | 5 months
  To collect data to improve the performance of the NOL algorithm in the study population
Efficacy outcome | 10 months
  The ability of the NOL index to discriminate between periods of painful and non-painful periods

SECONDARY OUTCOMES:
Efficacy outcome | 10 months
  NOL-index performance to detect pain in comparison to PAINAD, BPS pain scores

CONTACTS AND LOCATIONS:
Overall Officials: Adi Sasson, Dr., Principal Investigator — DOROT, Netanya Geriatric Medical Center
Locations (1):
- Dorot Netanya Gariatric Medical Center, Netanya, Israel

IPD SHARING:
Plan to Share IPD: No